CLINICAL TRIAL: NCT03914183
Title: Can a montméd Coloured Pen Needle (mCPN) Intervention Improve Injection Site Rotation Habits in Established Insulin Users
Brief Title: Can mCPN Intervention Improve Injection Site Rotation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pink Pearls Inc (Other)
Collaborators: Montméd (Unknown)
Responsible Party: Principal Investigator, Lori Berard, Nurse Consultant, Pink Pearls Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: mCPN
Record Dates: First submitted 2019-04-08; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Injection Site Rotation; Diabete Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Open label randomized control study of control (current standard of care) versus mCPN intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Standard of care arm - using insulin pen needles as previously prescribed
  Interventions: Device: Control
- mCPN intervention (Active Comparator): Each box of montméd Coloured Pen Needles (mCPN) has the following five features:
  i. Distinctively coloured pen needles ii. A user-defined association tool which is intended to help the patient associate each colour to a specific injection zone iii. A concise and intuitive educational message "Change color, change site" siteTM" iv. Unique packaging with educational content v. Four distinctive message-in-a-box educational sound-chips which serve to reinforce the recommended educational message on site rotation at home and come on every tenth time the pen needle box is opened The current research study has accordingly been designed to determine if a "pharmacist-dispensed montméd Coloured Pen Needle (mCPN) intervention" will improve injection site rotation relative to the standard dispensing of non-mCPN insulin pen needles.
  Interventions: Device: mCPN Intervention

INTERVENTIONS:
Device: mCPN Intervention — Each box of montméd Coloured Pen Needles (mCPN) has the following five features:
  i. Distinctively coloured pen needles ii. A user-defined association tool which is intended to help the patient associate each colour to a specific injection zone iii. A concise and intuitive educational message "Change color, change site" siteTM" iv. Unique packaging with educational content v. Four distinctive message-in-a-box educational sound-chips which serve to reinforce the recommended educational message on site rotation at home and come on every tenth time the pen needle box is opened
  Arms: mCPN intervention
Device: Control — Use of standard of care insulin pen needle
  Arms: Control

SUMMARY:
The current research study has accordingly been designed to determine if a "pharmacist-dispensed montméd Coloured Pen Needle (mCPN) intervention" will improve injection site rotation relative to the standard dispensing of non-mCPN insulin pen needles.

DETAILED DESCRIPTION:
Study Design and Conduct This is a 30-day, two-arm, randomized, controlled study.

Enrolled participants will be randomly assigned to one of the following study arms:

* Control group: participating pharmacists will dispense boxes of standard insulin pen needles to the patient participants
* mCPN group: participating pharmacists will dispense boxes of montméd Coloured Pen Needles to the patient participants

Study Sites and Participating Pharmacists All pharmacies in Canada that provide services to individuals with diabetes who use injectable insulin therapy will be eligible to participate in this study. All participating pharmacists who will play an active role in participant enrollment and the follow-up visits will be required to complete a participation consent form and 2 surveys. The first (Pre-study survey) should be completed after they have been fully trained on the study protocol and their study obligations, and before commencement of study enrollment. The second (Post-study survey) should be completed after the last patient has completed the 30-day follow-up visit. (Refer to Section 11 for the Study Flow).

Randomization Process Participating pharmacists will dispense one of the two study pen needles according to a computer-generated list that will be provided to the participating pharmacy upon site activation

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus or type 2 diabetes mellitus who have been using daily insulin therapy for 1 year or more
* Able to read the English text on the boxes of the pen needles

Exclusion Criteria:

* Individuals currently treated with a glucagon-like peptide 1 receptor agonist (GLP-1RA)
* Current or previous user of mCPN
* Individuals who are unable to understand or communicate in English
* Pregnant women
* Individuals with serious mental illnesses eg. dementia, schizophrenia disorders, bipolar disorders, major depression, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
The percentage of participants in the mCPN group who demonstrate an improvement (vs baseline performance) in the recommended site rotation techniques relative to the proportion of that in the control group. | 30 - 45 days

SECONDARY OUTCOMES:
Does a retail pharmacy-based, pharmacist-led mCPN intervention improve the knowledge base of pharmacists around injection site rotation | Study duration. 30 to 90 days
  The change the level of knowledge about the importance of site rotation as (importance scale) as measured by a 5 point likert scale; Unimportant (1) Slightly Important (2) Neither (3) Slightly Important (4) Very Important (5)
Does a retail pharmacy-based, pharmacist-led mCPN intervention increase confidence in providing injection site rotation counselling | Study duration 30 to 90 days
  The change in the level of confidence in providing injection site rotation counselling (Confidence Scale) using a 5 point likert scale: Not confident (1) Little Confidence (2)Neither (3) Somewhat Confident (4) Very confident (5)
increase/change in injection zone size | 30-45 days
  Assessment of injection rotation from pre to post survey patient reported
percentage of participating patients who change their needles more often (patient reported), | 30 - 45 days
  Assessment of needle reuse or lack of reuse from pre to post survey patient reported
the percentage of participating patients who decide to continue using mCPN upon study completion | 30- 45 days
  Willingness to continue with intervention needle from post survey - patient reported

CONTACTS AND LOCATIONS:
Overall Officials: Lori Berard, Principal Investigator — Pink Pearls Inc
Locations (14):
- Canada (14):
  - Shoppers Drug Mart 2335, Calgary, Alberta
  - Claresholm Pharamcy, Claresholm, Alberta
  - Rexall 7236, Edmonton, Alberta
  - Shoppers Drug Mart 2401, Okotoks, Alberta
  - Kipp Mallery Pharmacy, Kamloops, British Columbia
  - Our Own Health Centre, Winnipeg, Manitoba
  - Shoppers Drug Mart 535, Winnipeg, Manitoba
  - Kennegecasis Drugs, Rothesay, New Brunswick
  - Zak's Pharmacy, Milton, Ontario
  - Niagara Pharmacy, Niagara Falls, Ontario
  - Northgate Pharmacy, Sarnia, Ontario
  - Murphy's Cornwall Pharmacy, Cornwall, Prince Edward Island
  - Pharmacie Jacques Bourget PJC076, Laval, Quebec
  - Pharmacy Jean-Coutu Raffaele Delli Colli & Gino Consolante, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-07-23): https://cdn.clinicaltrials.gov/large-docs/83/NCT03914183/Prot_SAP_ICF_000.pdf